CLINICAL TRIAL: NCT00856869
Title: A Study in Healthy Volunteers and Patients With Liver Cirrhosis and Non-Alcoholic Steatohepatitis (NASH) to Assess the Effects of Age, Gender, Chronic Liver Disease, and Prandial Effects on the Clearance of Cholyl-Lysyl-Fluorescein (NRL972) an an in-Vivo Marker of Liver Function in Man.
Brief Title: Clearance of NRL972 in Patients With Cirrhosis, Nonalcoholic Steatohepatitis (NASH) and in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Vice President Clinical Development, Norgine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NRL972-02/2003(ACPS)
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2009-03

CONDITIONS: Hepatic Cirrhosis; Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Liver Cirrhosis; Non-alcoholic Fatty Liver Disease | interventions — NRL972

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- 1 YM (Experimental): Healthy young males
  Interventions: Drug: NRL972
- 2 EM (Experimental): Healthy elderly males
  Interventions: Drug: NRL972
- 3 YF (Experimental): Healthy young females
  Interventions: Drug: NRL972
- 4 EF (Experimental): Healthy elderly females
  Interventions: Drug: NRL972
- 5 NASH (Experimental): Patients with presumed NASH
  Interventions: Drug: NRL972
- 6 CTP-A (Experimental): Patients with hepatic cirrhosis CTP-class A
  Interventions: Drug: NRL972
- 7 CTP-BC (Experimental): Patients with hepatic cirrhosis CTP-class B and C
  Interventions: Drug: NRL972

INTERVENTIONS:
Drug: NRL972 — Single 2 mg intravenous injection administered once after an overnight fast and once after a standard meal
  Arms: 1 YM
Drug: NRL972 — Single 2 mg intravenous injection administered once after an overnight fast and once after a standard meal
  Arms: 2 EM
Drug: NRL972 — Single 2 mg intravenous injection administered once after an overnight fast and once after a standard meal
  Arms: 3 YF
Drug: NRL972 — Single 2 mg intravenous injection administered once after an overnight fast and once after a standard meal
  Arms: 4 EF
Drug: NRL972 — Single 2 mg intravenous injection administered once after an overnight fast and once after a standard meal
  Arms: 5 NASH
Drug: NRL972 — Single 2 mg intravenous injection administered once after an overnight fast and once after a standard meal
  Arms: 6 CTP-A
Drug: NRL972 — Single 2 mg intravenous injection administered once after an overnight fast and once after a standard meal
  Arms: 7 CTP-BC

SUMMARY:
The study was conducted to describe and compare the plasma pharmacokinetics of NRL972 administered after a standard meal and while fasted in patients with hepatic cirrhosis (Child-Turcotte-Pugh [CTP] class A-C), NASH, young and elderly healthy males, and young and elderly healthy females, to assess the effects of liver dysfunction, gender, age and prandial intestinal hyperaemia on the clearance of NRL972. In addition, the study was to provide information on the safety and tolerability of repeated intravenous doses of NRL972 in these populations.

ELIGIBILITY:
Inclusion Criteria:

General - all subjects

1. Males or females (females of non-childbearing potential or of childbearing potential while taking medically appropriate contraception)
2. Caucasian
3. BMI: between 19 and 34 kg.m-2
4. BW: between 45 and 110 kg
5. willing and able to provide informed consent Healthy volunteers (group N)
6. Age: 18 - 40 years (inclusive) e.g. > 60 years
7. Assessed as healthy based on the pre study examination Hepatic cirrhosis
8. Age: 18 - 75 years
9. stable compensated liver cirrhosis (cryptogenic, posthepatic, alcoholic) with histo-logical or macroscopic (e.g. laparascopy, biopsy, ultrasound sonography or other adequate imaging techniques) confirmation Nonalcoholic steatohepatitis (NASH)
10. Age: 18 - 75 years
11. Diagnosis of NASH confirmed by liver biopsy

Exclusion Criteria:

General - all subjects

1. Previous participation in the trial
2. Participant in any other trial during the last 90 days
3. Donation of blood during the last 60 days or a history of blood loss exceeding 450 mL within the last 3 months
4. History of any clinically relevant allergy
5. Uncontrolled diabetes mellitus or any further intolerability of the Galactose test
6. Presence of acute or chronic infection
7. Resting systolic blood pressure > 160 or < 90 mmHg, diastolic blood pressure > 95 or < 50 mmHg
8. Clinically relevant ECG-abnormalities, prolonged QTc with > 450 msec in males and > 460 msec in females in particular
9. Clinically relevant ECG-abnormalities that constitute a contraindication for the Lido-cain-MEG'-X-test
10. Positive HIV test
11. Positive alcohol or urine drug test on recruitment
12. Daily use of > 30 gr alcohol
13. Smoking more than 15 cigarettes/day or equivalent of other tobacco products
14. Use of prohibited medication
15. Suspicion or evidence that the subject is not trustworthy and reliable
16. Suspicion or evidence that the subject is not able to make a free consent or to under-stand the information in this regard

    General - all females
17. Positive pregnancy test
18. Lactating
19. Not using appropriate contraception in premenopausal women All healthy subjects
20. Presence or history of any relevant comorbidity (list of past and present diseases will be reviewed by an expert panel)
21. Presence of any relevant abnormality in the laboratory safety tests, especially low haemoglobin, increased liver enzymes, reduced serum creatinine (laboratory test abnormalities will be reviewed by an expert panel)
22. Positive serology for HBsAg, anti HBc and anti HCV
23. History of alcohol and/or drug abuse.

    Patients with hepatic disease
24. Biliary liver cirrhosis
25. Liver impairment due to space-occupying processes (e.g. carcinoma)
26. State after liver transplantation or patient scheduled for liver transplantation
27. Fluctuating or rapidly deteriorating hepatic function
28. Significant bleeding diathesis
29. Oesophageal bleeding within the last 8 weeks before study entry
30. Ascites > 6 L on abdominal US
31. Number Connection test: time to connect 25 consecutive numbers > 30 sec
32. Presence or history of any relevant comorbidity other than hepatic disease (list of past and present diseases will be reviewed by an expert panel)
33. Clinically relevant abnormal laboratory values other than those associated or sufficiently explained by the existing liver disease (laboratory test abnormalities will be reviewed by an expert panel)
34. History of drug or alcohol abuse within 2 months prior to dosing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-08; Primary Completion 2005-02 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Clearance of NRL972 after a standard meal and while fasted in healthy volunteers, patients with NASH and patients with hepatic cirrhosis. | Up to 4 hours post administration of NRL972

SECONDARY OUTCOMES:
Adverse events and changes in physical findings from baseline | Up to 4 hours post-dosing
Effects of vital signs: blood pressure, pulse rate | Up to 4 hours post-dosing
Effects on electrocardiogram | Up to 4 hours post-dosing
Changes in haematology, clinical chemistry, urinalysis | Up to 4 hours post-dosing

CONTACTS AND LOCATIONS:
Overall Officials: Zahariy Krastev, MD, Principal Investigator — St. Ivan Rilski's University Hospital; Hans-Jürgen Gruss, MD, Study Director — Norgine
Locations (1):
- UMHAPT St. Ivan Rilski's University Hospital, Sofia, Bulgaria